CLINICAL TRIAL: NCT01511913
Title: A Multi-National, Prospective, Observational Study in Patients With Unresectable or Metastatic Melanoma
Acronym: IMAGE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-143; ENCEPP/SDPP/2723 (Other: Euro. Ntwk. of Ctrs. for Pharmacoepidemiology and Pharmacovigilance)
Record Dates: First submitted 2011-11-15; First posted 2012-01-19 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Advanced Cutaneous Melanoma
Keywords: Unresectable or metastatic cutaneous melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ipilimumab treatment cohort of 1106 prospective participants
- Non-Ipilimumab treatment cohort of 305 prospective participants
- Retrospective cohort of 177 participants

SUMMARY:
The purpose of this study is to examine the safety of Ipilimumab and patterns of use in the treatment of unresectable or metastatic melanoma in the post-approval setting

DETAILED DESCRIPTION:
Time Perspective: this study does have a retrospective component involving a subset of patients

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Diagnosis of unresectable or metastatic melanoma
* Age of 18 years or older at time of entry into the study
* Patients who have initiated treatment for unresectable or metastatic melanoma at medical practice (e.g. community-based, office-based, hospital-based, academic setting)within 21 days before informed consent for this study OR in the case where treatment has not yet been initiated, documentation that the treatment strategy was determined before informed consent for this study, and treatment must be initiated within 28 days after informed consent
* Ipilimumab-treated patients must be receiving treatment for the indication(s) approved in their country of residence or where they are receiving treatment

Exclusion Criteria:

* Current or pending participation in a clinical trial examining therapy for the treatment of any cancer (including unresectable or metastatic melanoma)
* Current use of therapy to treat a primary cancer other than melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be selected from approximately 200 medical practice sites (e.g. community-based, office-based, hospital-based, academic setting) in several European Union countries, Central America, North America, and South America, as well as Australia and Israel.
Sampling Method: Non-Probability Sample
Enrollment: 1411 (Actual)
Dates: Start 2012-06-03 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse reactions in patients treated with Ipilimumab in the post-approval setting | Every 12 months up to 5 years
Incidence rate with person-year-exposure and frequency estimate of adverse events/serious adverse events | Every 12 months up to 5 years
Frequency at which immunosuppressive therapy was administered to patients to manage treatment-related adverse events associated with Ipilimumab | Every 12 months up to 5 years
Patterns of disease monitoring as observed in a real-world setting | Every 12 months up to 5 years
  To evaluate patterns of care, descriptive statistics will describe treatment, dosing, regimen, indication, treatment rationales, management of treatment-related adverse events, reasons for treatment termination

SECONDARY OUTCOMES:
Quality of life (QoL), impact on work productivity, and overall satisfaction among patients receiving any therapy for unresectable or metastatic melanoma | Every 12 months up to 5 years
Resource utilization associated with advanced melanoma treatment | Every 12 months up to 5 years
  Descriptive statistics will be reported for healthcare utilization (inpatient, outpatient, emergency department and other ancillary services) and imputed costs
Overall survival (OS) in patients receiving Ipilimumab or other therapies for unresectable or metastatic melanoma | Every 12 months up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (174):
- United States (24):
  - Local Institution, Gilbert, Arizona
  - Local Institution, Hot Springs, Arkansas
  - Local Institution, Encinitas, California
  - Local Institution, La Jolla, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Denver, Colorado
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Lakeland, Florida
  - Local Institution, Miami Beach, Florida
  - Local Institution, Orange Park, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Niles, Illinois
  - Local Institution, Detroit, Michigan
  - Local Institution, Hattiesburg, Mississippi
  - Local Institution, Lincoln, Nebraska
  - Local Institution, Morristown, New Jersey
  - Local Institution, Canton, Ohio
  - Mid Ohio Onc/Hem, Inc, Columbus, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Middletown, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Everett, Washington
- Argentina (4):
  - Local Institution, CABA
  - Local Institution, Córdoba
  - Local Institution, Rosario- Santa Fe
  - Local Institution, San Miguel de Tucumán
- Australia (16):
  - Local Institution, Canberra, Australian Capital Territory
  - Local Institution, Corrimal, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, Port Macquarie, New South Wales
  - Local Institution, Tamworth, New South Wales
  - Local Institution, Tweeds Head, New South Wales
  - Local Institution, Wagga Wagga, New South Wales
  - Local Institution, Waratah, New South Wales
  - Local Institution, Cairns, Queensland
  - Local Institution, Douglas, Queensland
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Kurralta Park, South Australia
  - Local Institution, Frankston, Victoria
  - Local Institution, Malvern, Victoria
- Austria (6):
  - Local Institution, Feldkirch
  - Local Institution, Graz
  - Local Institution, Linz
  - Local Institution, Salzburg
  - Local Institution, Sankt Pölten
  - Local Institution, Vienna
- Belgium (7):
  - Local Institution, Brasschaat
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Haint Saint Paul
  - Local Institution, Hasselt
  - Local Institution, Kortrijk
  - Local Institution, Leuven
- Canada (7):
  - Local Institution, Moncton, New Brunswick
  - Local Institution, London, Ontario
  - Local Institution, Mississauga, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Québec, Quebec
  - Local Institution, Saskatoon, Saskatchewan
  - Local Institution, Québec
- France (19):
  - Local Institution, Bayonne
  - Local Institution, Besançon
  - Local Institution, Boulogne
  - Local Institution, Boulogne-sur-Mer
  - Local Institution, Brest
  - Local Institution, Clermont Ferrand Cédex 1
  - Local Institution, Dijon
  - Local Institution, Grenoble Cédex
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Montauban
  - Local Institution, Mougins
  - Local Institution, Nouvelle Caledonie
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Quimper
  - Local Institution, Soissons
  - Local Institution, Strasbourg
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (30):
  - Local Institution, Augsburg
  - Local Institution, Bochum
  - Local Institution, Buxtehude
  - Local Institution, Chemnitz
  - Local Institution, Darmstadt
  - Local Institution, Dessau-Roblau
  - Local Institution, Dortmund
  - Local Institution, Dresden
  - Local Institution, Düsseldorf
  - Local Institution, Frankfurt
  - Local Institution, Gera
  - Local Institution, Halle
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Jena
  - Local Institution, Koblenz
  - Local Institution, Lüdenscheid
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Marburg
  - Local Institution, Münster
  - Local Institution, Plauen
  - Local Institution, Quedlinburg
  - Local Institution, Recklinghausen
  - Local Institution, Rostock
  - Local Institution, Schwäbisch Hall
  - Local Institution, Stuttgart
  - Local Institution, Tübingen
  - Local Institution, Würzburg
- Greece (9):
  - Local Institution, Cholargós, Athens
  - Local institution, Goudi, Athens
  - Local Institution, Neo Faliro, Athens
  - Local Institution, Heraklion, Crete
  - Local Institution, Neas Efkarpia, Thessaloniki
  - Local Institutio, Alexandroupoli
  - Local Institution, Athens
  - Local Institution, Mezourlo
  - Local Institution, Neo Faliro
- Ireland (5):
  - Local Institution, Wilton, CORK
  - Local Institution, Cork
  - Local Institution, Dublin
  - Local Institution, Galway
  - Local Institution, Tullamore
- Israel (3):
  - Local Institution, Haifa
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
- Poland (4):
  - Local Institution, Bydgoszcz
  - Local Institution, Lodz
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Spain (14):
  - Local Institution, Barcelona
  - Local Institution, Donostia / San Sebastian
  - Local Institution, Las Palmas de Gran Canaria
  - Local Institution, Madrid
  - Local Institution, Palma
  - Local Institution, Palma de Mallorca
  - Local Institution, Pamplona
  - Local Institution, Santa Cruz de Tenerife
  - Local Institution, Santander
  - Local Institution, Santiago de Compostela; A Coruña
  - Local Institution, Seville
  - Local Institution, Terrassa
  - Local Institution, Valladolid
  - Local Institution, Zaragoza
- Switzerland (3):
  - Local Institution, Baden
  - Local Institution, Lugano
  - Local Institution, Zurich
- United Kingdom (23):
  - Local Institution, Rhyl, Denbigshire
  - Local Institution, London, England
  - Local Institution, Chelmsford, Essex, Essex
  - Local Institution, Southend, Essex
  - Local Institution, Belfast, Ireland
  - Local Institution, Cardiff, South Glamorgan
  - Local Institution, Birmingham
  - Local Institution, Bristol
  - Local Institution, Exeter
  - Local Institution, Hull
  - Local Institution, Leeds
  - Local Institution, Lincoln
  - Local Institution, London
  - Local Institution, Metropolitan Borough of Wirral
  - Local Institution, Oxfordshire
  - Local Institution, Plymouth
  - Local Institution, Poole
  - Local Institution, Preston
  - Local Institution, Staffordshire
  - Local Institution, Taunton, Somerset
  - Local Institution, Truro, Cornwall
  - Local Institution, Wolverhampton
  - Local Institution, Yeovil, Somerset

REFERENCES:
- [Result] Dalle S, Mortier L, Corrie P, Lotem M, Board R, Arance AM, Meiss F, Terheyden P, Gutzmer R, Buysse B, Oh K, Brokaw J, Le TK, Mathias SD, Scotto J, Lord-Bessen J, Moshyk A, Kotapati S, Middleton MR. Long-term real-world experience with ipilimumab and non-ipilimumab therapies in advanced melanoma: the IMAGE study. BMC Cancer. 2021 May 29;21(1):642. doi: 10.1186/s12885-021-08032-y. PMID 34051732
- [Result] Middleton MR, Dalle S, Claveau J, Mut P, Hallmeyer S, Plantin P, Highley M, Kotapati S, Le TK, Brokaw J, Abernethy AP. Real-world treatment practice in patients with advanced melanoma in the era before ipilimumab: results from the IMAGE study. Cancer Med. 2016 Jul;5(7):1436-43. doi: 10.1002/cam4.717. Epub 2016 Apr 26. PMID 27118102
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome